CLINICAL TRIAL: NCT03223168
Title: Noninvasive Negative Pressure Ventilation to Support Failing Fontan Physiology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, David Peng, Assistant Professor of Pediatrics and Communicable Diseases, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: HUM00131186
Record Dates: First submitted 2017-07-17; First posted 2017-07-21 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Failing Fontan Physiology; Pediatric Congenital Heart Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Hayek RTX ventilator (Experimental): Participants will receive noninvasive negative pressure ventilation.
  Interventions: Device: Hayek RTX ventilator

INTERVENTIONS:
Device: Hayek RTX ventilator — Participants will receive Noninvasive negative pressure from the Hayek RTX ventilator for 30 minutes during diagnostic catheterization procedure.

SUMMARY:
The purpose of this study is to assess for acute hemodynamic changes after implementation of noninvasive negative pressure ventilation (as compared with spontaneous respiration) in pediatric patients with Fontan failure using modern negative pressure ventilators

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Fontan physiology with clinical evidence of Fontan failure as defined by those with one of the following in addition to Fontan circulation: New York Heart Association Class II, fluid retention, cyanosis, protein losing enteropathy, renal/hepatic dysfunction and/or subjectively qualify for hemodynamic assessment (by primary cardiologist).

Exclusion Criteria:

1. Patients which will likely require intubation for catheterization
2. Severely depressed systemic ventricular systolic function
3. Baseline airway obstruction
4. Plastic bronchitis
5. Significant OUTFLOW obstruction

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2018-06-13 (Actual); Study Completion 2018-07-19 (Actual)

PRIMARY OUTCOMES:
Hemodynamics as characterized by change in pulmonary artery pressure | Baseline, 45 Minutes
  Pulmonary artery wedge pressure will be measured in millimeters of mercury (mmHg) at baseline and completion of noninvasive negative pressure ventilation.
Hemodynamics as characterized by change in pulmonary blood flow | Baseline, 45 Minutes
  Change in pulmonary blood flow will be measured at baseline and completion of noninvasive negative pressure ventilation.
Hemodynamics as characterized by change in systemic arterial saturation | Baseline, 45 Minutes
  Systemic arterial saturation measures the amount of oxygen in the blood stream. Systemic arterial saturation will be registered at baseline and completion of noninvasive negative pressure ventilation.
Hemodynamics as characterized by change in cardiac output | Baseline, 45 Minutes
  Cardiac output will be measured in liters per minute at baseline and completion of noninvasive negative pressure ventilation

CONTACTS AND LOCATIONS:
Overall Officials: David Peng, MD, Principal Investigator — University of Michigan
Locations (1):
- University of MIchigan, Ann Arbor, Michigan, United States